CLINICAL TRIAL: NCT06303596
Title: Investigating the Efficacy of Hippotherapy Program on Disease Symptoms, Quality of Life, Anxiety and Loneliness Levels in Patients With Schizophrenia: A Randomized Controlled Trial
Brief Title: Hippotherapy in Patients With Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hippotherapy in Schizophrenia
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Equine-Assisted Therapy; Schizophrenia
Keywords: hippotherapy; schizophrenia; quality of life; anxiety; loneliness
MeSH Terms: conditions — Schizophrenia; Anxiety Disorders | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator who collects the data is blinded to the allocation of groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental group (Experimental): The experimental group would receive standard psychiatric treatment.
  Additionally, the experimental group would be provided with a 16-session hippotherapy program for 8 weeks, as an adjuvant to standard psychiatric treatment.
  Interventions: Other: Hippotherapy; Other: Standard psychiatric treatment
- Other: Control group (Other): The control group would receive only standard psychiatric treatment.
  Interventions: Other: Standard psychiatric treatment

INTERVENTIONS:
Other: Hippotherapy — Hippotherapy: Hippotherapy in psychiatry is not concerned only about the patient sitting on a horse and the horseback movement influencing the physical condition of the patient and his functional and postural disorders. This therapy is concerned with positive effects on a patient's mental state and use mainly contact with the horse, work with the horse from the ground and riding on horseback. It aims for enjoyment, social communication, and the development of cognitive and executive functions.
  Arms: Experimental: Experimental group
Other: Standard psychiatric treatment — Standard psychiatric treatment: Standard psychiatric treatment includes medication and routine activities provided by the Community Mental Health Center.

SUMMARY:
This study will determine the efficacy of hippotherapy (horseback-riding) program, as an adjuvant to standard psychiatric treatment, on the outcomes of patients with schizophrenia. A randomized controlled trial is conducted in a Community Mental Health Center. All participants are randomized into two groups (experimental and control groups) using blocked randomization. All participants received the standard psychiatric treatment, while the experimental group is additionally provided with a 16-session hippotherapy program for 8 weeks. All participants will be evaluated using the Positive and Negative Syndrome Scale, State-Trait Anxiety Inventory, Quality of Life Scale, UCLA Loneliness Scale at both baseline and after the intervention.

DETAILED DESCRIPTION:
Background: Schizophrenia is a multifactorial disorder characterized by cognitive and affective symptoms such as distortions of thinking and perception and loss of normal affective expressiveness. Since schizophrenia is a complex disorder, the management of the disease should include a combination of medication, psychotherapy and other supportive psychosocial interventions. One of the commonly used psychosocial interventions is hippotherapy which is incorporated into comprehensive rehabilitation therapy sessions aimed at restoring lost function, alleviate, minimize or eliminate physical, psychological, social or mental disability of the patients with various disorders.

Aim: The investigators hypothesize that hippotherapy, as an adjuvant to standard psychiatric treatment, could have significant effect on disease symptoms, quality of life, anxiety and loneliness levels of patients with schizophrenia. Therefore, in this study, the investigators will determine the effect of hippotherapy on disease symptoms, quality of life, anxiety and loneliness levels in patients with schizophrenia.

Methods: The study is designed as a single-blinded, randomized controlled trial. The sample of this study will be selected from patients who are eligible for the study and registered at the Community Mental Health Center. These centers aiming to increase the functional and mental recovery of patients with schizophrenia are composed of a team where different professionals as psychiatrists, psychologists, social workers, and nurses are present. In these centers, there are activities aimed at providing skills in business and social areas, training groups for disease, and giving information on medication and disease management. Participants are randomly allocated into two groups using blocked randomization. All participants received the standard psychiatric treatment, while the experimental groups are additionally provided with a 16-session hippotherapy program for 8 weeks.

Participants and demographic data: Participants who have been diagnosed with schizophrenia take part in the study after informed consent is obtained. The participants are able to express themselves and to individually complete the Positive and Negative Syndrome Scale, State-Trait Anxiety Inventory, Quality of Life Scale, UCLA Loneliness Scale.

Measures: The demographic characteristics, including variables such as sex, age, duration of disease, years of education, marital status, work status, and medications, will be recorded. In addition, four scales will be administered to patients for evaluating disease symptoms, quality of life, anxiety and loneliness levels.

Procedure and Data collection: Ethical approval is obtained from the Local Medical Ethics Committee. Following informed consent, each participant will fill out a demographic questionnaire and complete the Positive and Negative Syndrome Scale, State-Trait Anxiety Inventory, Quality of Life Scale, UCLA Loneliness Scale at baseline and after the intervention. A well-trained and licensed psychiatric nurse will perform the data collection and assists the participants if there were difficulties reading or understanding the questionnaires.

Statistical analysis: This study will employ Statistical Package for Social Sciences (SPSS) Version 26.0 to analyze the collected data. The data analyses will include demographic variables and the scores of the Positive and Negative Syndrome Scale, State-Trait Anxiety Inventory, Quality of Life Scale, UCLA Loneliness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with schizophrenia,
* Being at an age of older than 18 years,
* Being registered with and treated at the Community Mental Health Center,
* Being at remission period (a stable condition) at the time of enrollment and throughout the study.
* Being able to provide written informed consent and comprehend the instruments.

Exclusion Criteria:

* The participants who suffer from other comorbid psychiatric disorders (depression, personality disorder, substance addiction, etc.),
* The participants who are not willing to sign the consent.
* The participants who have physical health problems that would prevent horseback-riding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | For two study groups: at pre-intervention and immediately after the intervention.
  The Positive and Negative Syndrome Scale is used for measuring symptom severity of schizophrenia. The PANSS is a 30-item clinician-administered rating scale. It quantifies positive symptoms, which refer to an excess or distortion of normal functions (e.g., hallucinations and delusions), and negative symptoms, which represent a diminution or loss of normal functions.
State-Trait Anxiety Inventory (STAI) | For two study groups: at pre-intervention and immediately after the intervention.
  The STAI is a self-report scale that assesses separate dimensions of "state" and "trait" anxiety. Examples of what the STAI measures include feelings of apprehension, tension, nervousness, and worry.
The Quality of Life Scale (QLS) | For two study groups: at pre-intervention and immediately after the intervention.
  The Quality of Life Scale (QLS) is a 21-item scale rated from a semi-structured interview providing information on symptoms and functioning. It is divided into four dimensions: Intrapsychic Foundations, Interpersonal Relations, Instrumental Role Functioning, and Common Objects and Activities. The total score of the scale and each of the domains ranges from 0 to 6.
UCLA Loneliness Scale | For two study groups: at pre-intervention and immediately after the intervention.
  UCLA Loneliness Scale is a 20-item scale which designed to measure one's subjective feelings of loneliness as well as feelings of social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Oztürk, Ph.D., Assist. Prof., Study Director — Erzurum Technical University; Nurgül Karakurt, Ph.D., Assist. Prof., Principal Investigator — Erzurum Technical University; Elif O Tozoğlu, M.D., Principal Investigator — Erzurum Community Mental Health Center; Musa Eymir, Ph.D., PT, Assist. Prof., Principal Investigator — Erzurum Technical University; Serdar Ulusoy, Principal Investigator — Ataturk University
Locations (1):
- Erzurum Technical University, Erzurum Community Mental Health Center, Erzurum, Turkey (Türkiye)